CLINICAL TRIAL: NCT02234492
Title: The Effects of Statin Therapy on Coronary Flow Reserve and Inflammatory Markers in HIV-Positive Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Ontario HIV Treatment Network (Network)
Responsible Party: Principal Investigator, Gary Small, Associate Professor in Cardiology and Clinician Investigator, Ottawa Heart Institute Research Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20140263-01H
Record Dates: First submitted 2014-08-20; First posted 2014-09-09 (Estimated); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Human Immunodeficiency Virus (HIV); Cardiovascular Disease (CVD)
Keywords: Human immunodeficiency virus (HIV); Statin therapy; Cardiovascular disease (CVD); Coronary Flow Reserve (CFR); Positron Emission Tomography (PET); Myocardial contrast echocardiography (MCE)
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Cardiovascular Diseases | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rosuvastatin (Active Comparator): Rosuvastatin 10mg once daily for 6 months.
  Interventions: Drug: Rosuvastatin
- No rosuvastatin (No Intervention): No rosuvastatin- this group will continue with their current medical therapy for 6 months.

INTERVENTIONS:
Drug: Rosuvastatin — Comparison of rosuvastatin to no rosuvastatin
  Other Names: Crestor
  Arms: Rosuvastatin

SUMMARY:
The purpose of this study is to determine whether the use of rosuvastatin in Human Immunodeficiency Virus (HIV) infected individuals lowers inflammation in blood vessels, improves blood circulation in the small arteries that provide nutrients to the heart muscle and improves neurocognitive function.

DETAILED DESCRIPTION:
HIV is a chronic inflammatory disease. Patients with HIV are at a high risk of cardiovascular disease (CVD) which may be related to this state of chronic inflammation. HIV infected individuals are at up to four times higher risk of suffering a heart attack (also know as acute coronary syndrome).

The medicine rosuvastatin, commonly used to treat high cholesterol, has been shown to reduce inflammation in arteries in the general population and also in patients with high risk for heart problems.

72 subjects with HIV infection will be enrolled and divided into 2 groups of 36.

Group 1: Treatment Group: Participants will receive a low dose of rosuvastatin, 10mg, for 6 months in addition to their current medical therapy.

Group 2: Control Group: Participants will not receive rosuvastatin for 6 months and will continue with their current medical therapy.

Participants in both groups will undergo blood tests, Myocardial Contrast Echocardiography (MCE) scan and a Positron Emission Tomography/Computed Tomography PET/CT scan using a radioactive tracer called fluorodeoxyglucose (FDG-PET), monocyte and serum cytokine studies at baseline and 6 months.

10 subjects without HIV will also be enrolled to undergo monocyte and serum cytokine blood tests only, for comparison.

ELIGIBILITY:
Inclusion Criteria:

* 40-90 years of age
* documented evidence of HIV infection
* on standard antiretroviral therapy(ART) for >1 years
* viral load persistently below the limits of detection while on ART
* current Cluster of Differentiation Antigen 4 (CD4) count >350 cells/microlitre
* baseline Framingham risk score of 10-20%

Exclusion Criteria:

* uncontrolled diabetes mellitus (glycated hemoglobin (HbA1C) >6.5% or fasting glucose >7.0 mmol/L)
* uncontrolled hypertension (systolic blood pressure >160 or diastolic blood pressure >90)
* known coronary artery disease (CAD) e.g. previous myocardial infarction, revascularization procedure, or history of angina
* chronic renal failure (glomerular filtration rate (GFR) <60 ml/min)
* total cholesterol >5.8 mmol/L
* Low-density lipoprotein (LDL) cholesterol >4.0 mmol/L
* already receiving a statin for baseline dyslipidemia
* pregnant or lactating
* active untreated Hepatitis B or C
* diagnosis or clinical evidence of a concomitant inﬂammatory/autoimmune disease
* patients at baseline demonstrating regional perfusion abnormalities (confined to individual coronary territories) following stress MCE will be excluded and further management will be according to local best practice guidelines

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-09; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Correlation between coronary flow reserve (CFR) and maximum target to background ratio (TBRmax). | At baseline
  At baseline, correlation between CFR by MCE and vascular inflammation (TBRmax) by FDG-PET/CT will be assessed. We anticipate good overall concurrence.

SECONDARY OUTCOMES:
Change in CFR | At 6 months
  Changes in CFR as measured by MCE will be evaluated over six months in HIV+ patients on ART and treated with rosuvastatin versus those not on a statin. Our study will be one of the first to examine the effects of rosuvastatin on measures of both inflammation and CFR in HIV+ patients.
Change in TBRmax. | At 6 months
  Changes in vascular inflammation (TBRmax) as measured by FDG-PET/CT will be evaluated over six months in HIV+ patients on ART and treated with rosuvastatin versus those not on a statin.
Change in neurocognitive function | At 6 months
  Changes in neurocognitve function as measured by a neuropsychological test battery (AMS-III Spatial Span, WAIS-R Digit Symbol, Hopkins Verbal Learning Test, Grooved Pegboard, Trail Making Tests A&B, Letter Numbering Sequencing , Patient's Assessment of Own Functioning, Center for Epidemiologic Studies-Depression Scale) will be evaluated over six months .

CONTACTS AND LOCATIONS:
Overall Officials: Girish Dwivedi, MD MRCP PhD, Study Director — University of Ottawa Heart Institute, Harry Perkins Institute of Medical Research; Gary Small, MD MRCP, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (2):
- Canada (2):
  - The Ottawa Hospital-General Campus, Ottawa, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No